CLINICAL TRIAL: NCT03594253
Title: Randomized Control Trial of Regulation Focused Psychotherapy for Children (RFP-C) With Externalizing Behaviors
Brief Title: Evaluation of Regulation Focused Psychotherapy for Children
Acronym: RFP-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeshiva University (Other)
Collaborators: The FAR Fund (Unknown)
Responsible Party: Principal Investigator, Tracy Prout, Assistant Professor, Yeshiva University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-6595
Record Dates: First submitted 2018-02-23; First posted 2018-07-20 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Oppositional Defiant Disorder; Oppositional Defiant Disorder in Children
Keywords: oppositional defiant disorder; regulation focused psychotherapy for children; emotion regulation; psychodynamic psychotherapy
MeSH Terms: conditions — Oppositional Defiant Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Regulation Focused Psychotherapy for Children (RFP-C; Hoffman & Rice with Prout, 2015) is a novel, manualized, time-limited psychodynamic treatment approach for children who manifest disruptive behaviors and emotional dysregulation. RFP-C conceptualizes children's externalizing behaviors as expressions of maladaptive defenses or impaired emotion regulation (ER). The child's behaviors are understood as products of developmental delays in implicit ER (Rice & Hoffman, 2014). Externalizing behaviors are conceptualized both as biologically-driven products and as functional attempts to defend against painful emotions by protecting the child from disturbing feelings such as sadness, shame, and guilt. This 16-session (plus four parent sessions) psychotherapy method iteratively addressing a child's disruptive behaviors as strategies to avoid painful affect. RFP-C is hypothesized to address developmental immaturity of the implicit ER system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFP-C (Experimental): Regulation Focused Psychotherapy for Children (RFP-C; Hoffman & Rice with Prout, 2015) is a novel, manualized, time-limited psychodynamic treatment approach for children who manifest disruptive behaviors and emotional dysregulation. Throughout the 16 sessions of play therapy and four parent meetings, the clinician works with the parents and the child to increase understanding that all behavior, even disruptive behavior, has meaning in the service of emotional and behavioral regulation. This insight leads to a decreased need and reliance to act on the distressing emotions (e.g. less need for disruptive behaviors) and an increased ability to tolerate, work through, and talk about the feelings that previously needed to be warded off.
  Interventions: Behavioral: Regulation Focused Psychotherapy for Children
- Wait List control (No Intervention): Participants assigned to this condition will receive no intervention. They may continue on current medication regimens (no major changes) but may not be enrolled in psychological treatments. They will be evaluated weekly via phone call with primary caregiver. At the conclusion of this 10-week wait list period all participants assigned to this condition will receive RFP-C treatment.

INTERVENTIONS:
Behavioral: Regulation Focused Psychotherapy for Children — RFP-C is a manualized, psychodynamic psychotherapy that last 10 weeks. Children meet individually with a therapist for play therapy (twice a week for 16 sessions) and parents meet with the therapist for four full sessions (without the child).
  Other Names: RFP-C
  Arms: RFP-C

SUMMARY:
The main objective of this project is to conduct a study of RFP-C for children with disruptive behaviors. Regulation Focused Psychotherapy for Children (RFP-C) is a twice a week, play therapy intervention.

DETAILED DESCRIPTION:
Background/Significance Currently, there are no empirically supported, manualized psychodynamic treatments for children and adolescents with disruptive behavior problems. Many barriers exist to providing effective treatment, including the large dropout rates in child psychotherapy, especially when multiple risk factors are present, such as maternal stress, greater symptom severity, and lower socioeconomic status. In order to remain viable and competitive, clinicians and researchers must demonstrate that psychodynamic approaches are valuable in terms of positive clinical outcomes, cost-effectiveness, and ease of implementation across a range of settings and disciplines.

Externalizing behaviors are common in a wide range of child mental health problems, including oppositional defiant disorder, disruptive mood dysregulation disorder, and conduct disorder. These behaviors have high prevalence rates, ranging from 15 to 34 percent. These problems frequently result in the referral of young children to mental health providers and they are costly to the healthcare system overall . The current approach to these types of problems is to provide behavioral parent management training (PMT) to parents of the child in distress. These programs include Parent-Child Interaction Therapy, Triple P-Positive Parenting Program, or The Incredible Years. Behavioral parent training programs are widely used because the evidence shows they are efficacious for children with externalizing behaviors. PMT relies on traditional cognitive behavioral strategies in working with the parent, including behavioral modeling, rewards, reinforcement, and punishment. The parent is taught to set limits for the child and to direct and to shape behavior. A significant limitation associated with behavioral parent programs (and psychotherapy with children and adolescents in general) is elevated attrition rates for vulnerable populations due to factors such as low socioeconomic status, ethnic minority status, parental functioning, maternal stress, low parental motivation, and child symptom severity. Parental attrition in behavioral parent training is also due to parental attribution about where the problem resides - within the child. PMT is directed at the parent, which contradicts the parent's understanding of the cause and nature of the problem, thus sometimes further reducing motivation to seek and complete treatment.

Regulation Focused Psychotherapy for Children (RFP-C) is a novel, manualized, time-limited psychodynamic treatment approach for children who manifest disruptive behaviors and emotional dysregulation. RFP-C conceptualizes children's externalizing behaviors as expressions of maladaptive defenses or impaired emotion regulation (ER). The child's behaviors are understood as products of developmental delays in implicit ER. This system has defined neurofunctional correlates which permit a targeting of the therapeutic work to brain-based deficits in the child's normative development. Externalizing behaviors are thus conceptualized both as biologically-driven products and as functional attempts to defend against painful emotions by protecting the child from disturbing feelings such as sadness, shame, and guilt. RFP-C relies heavily on the child being able to experience distressing affects through play and through the relationship with the therapist. Throughout the 16 sessions of play therapy and several parent meetings, the clinician works with the parents and the child to increase understanding that all behavior, even disruptive behavior, has meaning in the service of emotional and behavioral regulation. This insight leads to a decreased need and reliance to act on the distressing emotions (e.g. less need for disruptive behaviors) and an increased ability to tolerate, work through, and talk about the feelings that previously needed to be warded off.

This 16-session (plus four parent sessions) psychotherapy method operationalizes individual play therapy approaches for children with externalizing behaviors, including oppositional defiant disorder (ODD). Play therapy has long been the mainstay of community mental health with children and adolescents and has demonstrated efficacy, though no one has developed a play-based manualized treatment for children to date. Through iteratively addressing a child's disruptive behaviors as strategies to avoid painful affect, RFP-C is hypothesized to address developmental immaturity of the implicit ER system.

Rationale There is a critical need for the development, evaluation, and implementation of evidence-based psychodynamic treatments for children and adolescents. Regulation Focused Psychotherapy for Children is a novel, manualized, time-limited psychodynamic treatment approach for children who manifest disruptive behaviors and emotional dysregulation. To date, we have only conducted a small pilot study of the RFP-C method. No clinical trial has been conducted to determine the outcomes associated with RFP-C in a larger sample. The immediate objective of this proposal is to conduct a randomized controlled trial with 20 children in order to evaluate comparable efficacy to a waitlist control group.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing symptoms of ODD
* Fluent in English
* Not diagnosed with severe autism spectrum disorder
* Able to attend therapy twice a week for 10 weeks in the Bronx
* No concurrent therapy services (psychosocial groups and Individualized Education Plan supports are acceptable)

Exclusion Criteria:

* Active Administration for Children's Services (ACS)/Child Protective Services (CPS) involvement
* Severe autism spectrum disorder

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Oppositional Defiant Disorder Rating Scale | Pre and post treatment (prior to randomization, after 10 week wait list period if appropriate, and again after completion of 10 week treatment)
  symptom inventory based on Diagnostic and Statistical Manual (DSM) 5 - parent report Total possible score ranges from 0 - 24 with 0 representing no oppositional defiant disorder symptoms and 24 representing the most intense and frequent degree of oppositional defiant symptoms

SECONDARY OUTCOMES:
Emotion Regulation Checklist | Pre and post treatment (prior to randomization, after 10 week wait list period if appropriate, and again after completion of 10 week treatment)
  Parent report of ER capacities
  The ERC assessed children's ability to manage emotional experiences using a 24-item, four- point Likert scale (1 = Never, 4 = Always). The questionnaire yields two subscales: 1) adaptive emotion regulation (e.g. "Can modulate excitement in emotionally arousing situations", range 10-40 with higher scores representing more adaptive ER), which assesses situational appropriateness of affective displays, empathy and emotional self-awareness; and 2) lability/negativity (e.g. "Exhibits wide mood swings", range 14-56, with higher scores representing more lability/negativity), which assesses mood lability, lack of flexibility, dysregulated negative affect and inappropriate affective displays.
Emotional Regulation Questionnaire - Child & Adolescent | Pre and post treatment (prior to randomization, after 10 week wait list period if appropriate, and again after completion of 10 week treatment)
  Child report of ER capacities
  The questionnaire consists of 10 items capturing two specific emotion regulation strategies, cognitive reappraisal and expressive suppression on a 7-point Likert scale, where 1 means "strongly disagree", 4 "neutral", and 7 means "strongly agree". Higher mean score on a subscale indicates that the strategy is more endorsed. The cognitive reappraisal scale has 6 items and the expressive suppression has 4 items.
Child Behavior Checklist | Pre and post treatment (prior to randomization, after 10 week wait list period if appropriate, and again after completion of 10 week treatment)
  ODD subscale - six items on sub scale, scored by computer, reports T-scores; T-score below 60 is normal, 60-70 is borderline, >70 is clinical range

CONTACTS AND LOCATIONS:
Overall Officials: Tracy A. Prout, PhD, Principal Investigator — Ferkauf Graduate School of Psychology
Locations (1):
- Ferkauf Graduate School of Psychology - Yeshiva University, The Bronx, New York, United States

REFERENCES:
- [Derived] Prout TA, Rice T, Chung H, Gorokhovsky Y, Murphy S, Hoffman L. Randomized controlled trial of Regulation Focused Psychotherapy for children: A manualized psychodynamic treatment for externalizing behaviors. Psychother Res. 2022 Jun;32(5):555-570. doi: 10.1080/10503307.2021.1980626. Epub 2021 Sep 28. PMID 34583626
- See also: Study Website — https://www.centerforrfp.org/